CLINICAL TRIAL: NCT03836092
Title: Identification of AF Triggers, Initiators and Perpetuators by Electro Cardio-Graphic Imaging (ECGI) in Patients With Persistent Atrial Fibrillation
Brief Title: ECGI in Patients With Persistent Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Pacific Rim Electrophysiology Research Institute (Other)
Responsible Party: Principal Investigator, Koonlawee Nademanee, MD, Principal Investigator, Pacific Rim Electrophysiology Research Institute
Other Study IDs: PACIFICRERI3
Record Dates: First submitted 2019-01-27; First posted 2019-02-11 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Radiofrequency ablation — RF applications were delivered with a maximal temperature of 43°C at the catheter tip (SmartTouch Navistar Thermocool catheter) and at the power between 25-50 watts. The primary end points during RF ablation were either complete elimination of areas with CFAE or conversion of AF to normal sinus rhythm (SR). When areas with CFAE were completely eliminated but the atrial arrhythmias persisted (organized atrial flutter or atrial tachycardia), they were subsequently mapped and ablated (occasionally in conjunction with ibutilide, 1 - 2 mgs intravenously over 10 minutes).

SUMMARY:
To determine the values and limitations of ECGI in guiding ablation and risk stratification in patients with persistent atrial fibrillation.

DETAILED DESCRIPTION:
The patient population will include symptomatic persistent AF patients (N=50). The total of fifty patients will be studied to determine:

* The values and limitations of ECGI in identifying atrial fibrillation (AF) triggers, AF initiators and AF perpetuators as targets sites for catheter ablations in patients with persistent AF.
* The mechanisms of residual atrial tachycardia/flutter (Res-AT/AFl) after AF substrate ablations by targeting complex fractionated atrial electrograms (CFAE).
* If there is a relationship between primary CFAE sites and driver sites or other distinct patterns from the ECGI mapping system.
* The rate of AF termination to sinus rhythm after ablation at target sites identified by ECGI

ELIGIBILITY:
Inclusion Criteria:

* Patients are diagnosed as persistent AF. Persistent AF was defined as continuous AF from 7 days to 12 months and long- lasting AF beyond twelve months.
* Patients who are symptomatic
* Patients who are willing to sign consent and be followed post procedure in an out- patient arrhythmia clinic

Exclusion Criteria:

* Patients under 18 years or over 85 years of age.
* Patients with chronic alcoholism.
* Recent myocardial infarction within one month of the study.
* Significant debilitating diseases or a terminal disease.
* Patients with documented left atrial thrombus.
* Medical or mental conditions precluding a long-term follow-up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will include symptomatic persistent AF patients (N=50). The total of fifty patients will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Freedom from Atrial Fibrillation | 1 year
  termination via ablation from atrial fibrillation during follow up period

SECONDARY OUTCOMES:
termination via ablation from atrial fibrillation during procedure | over 6 months
  Termination of AF to NSR during procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Bumrungrad International Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nademanee K, McKenzie J, Kosar E, Schwab M, Sunsaneewitayakul B, Vasavakul T, Khunnawat C, Ngarmukos T. A new approach for catheter ablation of atrial fibrillation: mapping of the electrophysiologic substrate. J Am Coll Cardiol. 2004 Jun 2;43(11):2044-53. doi: 10.1016/j.jacc.2003.12.054. PMID 15172410
- [Result] Haissaguerre M, Hocini M, Denis A, Shah AJ, Komatsu Y, Yamashita S, Daly M, Amraoui S, Zellerhoff S, Picat MQ, Quotb A, Jesel L, Lim H, Ploux S, Bordachar P, Attuel G, Meillet V, Ritter P, Derval N, Sacher F, Bernus O, Cochet H, Jais P, Dubois R. Driver domains in persistent atrial fibrillation. Circulation. 2014 Aug 12;130(7):530-8. doi: 10.1161/CIRCULATIONAHA.113.005421. Epub 2014 Jul 15. PMID 25028391
- [Result] Conti S, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P, Verma A. Effect of Different Cutpoints for Defining Success Post-Catheter Ablation for Persistent Atrial Fibrillation: A Substudy of the STAR AF II Trial. JACC Clin Electrophysiol. 2017 May;3(5):522-523. doi: 10.1016/j.jacep.2016.12.006. Epub 2017 May 15. No abstract available. PMID 29759610
- [Result] Oketani N, Seitz J, Salazar M, Pisapia A, Kalifa J, Smit JJ, Nademanee K. Ablation of complex fractionated electrograms is useful for catheter ablation of persistent atrial fibrillation: Protagonist point of view. Heart Rhythm. 2016 Oct;13(10):2098-100. doi: 10.1016/j.hrthm.2016.06.036. Epub 2016 Jul 1. No abstract available. PMID 27374307
- [Result] Nademanee K, Amnueypol M, Lee F, Drew CM, Suwannasri W, Schwab MC, Veerakul G. Benefits and risks of catheter ablation in elderly patients with atrial fibrillation. Heart Rhythm. 2015 Jan;12(1):44-51. doi: 10.1016/j.hrthm.2014.09.049. Epub 2014 Oct 11. PMID 25257091